CLINICAL TRIAL: NCT00785746
Title: Improving Balance in Frail Elderly: A Randomized Clinical Trial of Two Methods to Enhance Strength (Stretch and Strength Versus Core Strength)
Brief Title: Improving Balance in Frail Elderly
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Nancy Mayo, BSc(PT), MSc, PhD, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SDR-06--010
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2010-03

CONDITIONS: Elderly; Frail
Keywords: elderly, balance, core, strength

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- core (Experimental): strength training of the core muscles.
  Interventions: Other: Core
- stretch and strength (No Intervention): This program consists of general stretching exercises and peripheral muscle strengthening exercises with a special emphasis on strengthening the upper extremity muscles because of their importance for ADL but not necessarily balance.

INTERVENTIONS:
Other: Core — We have devised a series of core strength training exercises that can be easily and safely performed under the supervision of trained staff. The exercises will be individualized depending on the participants' ability and health conditions. The majority, but not all, of exercises will be performed on or with exercise balls of different sizes and shapes, round for more advanced persons and oval for more frail persons.
  Arms: core

SUMMARY:
The objective of this pilot study is to estimate, for a frail elderly population, the extent to which balance improves following a Core-Strength training program in comparison to a Stretch & Strength program. A secondary objective is to explore the impact of core strength training on urinary incontinence.

DETAILED DESCRIPTION:
Participants will be randomized to one of the two exercise groups, Core-Strength training group or the Stretch & Strength group. The exercises will consist of 15-20 minute session for every day they attend the GDH. Measures will be made at admission, after 6 weeks of the program and at discharge if more than past 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* elderly persons attending the geriatric day hospital at the royal victoria hospital

Exclusion Criteria:

* persons who are not medically fit to participate in the Geriatric day hospital physiotherapy component.
* the individuals at high risk for falls

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | baseline, 6 weeks, discharge

SECONDARY OUTCOMES:
Functional walking capacity 6 minute walk test | baseline, 6 weeks, discharge
Gait speed | baseline, 6 weeks, discharge
Bridge Test | Baseline, 6 weeks, discharge
Activities-Specific Balance Confidence Scale (ABC Scale) | Baseline, 6 weeks, Discharge
International Consultation on Urinary Incontinence Questionnaire- Urinary Incontinence Short Form (ICIQ-UI) | Baseline, 6 weeks, discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Mayo, PhD, Principal Investigator — McGill University, Division of Clinical Epidemiology
Locations (1):
- McGill University-Royal Victoria Hospital Site, Montreal, Quebec, Canada